CLINICAL TRIAL: NCT02076841
Title: Tolerability and Quality of Life in Patients With Multiple Sclerosis Switched to Intramuscular Interferon Beta 1a Autoinjector (Avonex® PenTM)
Brief Title: Tolerability and Quality of Life Study in Participants Who Switched to Avonex Pen
Acronym: SFERA
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CHE-AVX-12-10348
Record Dates: First submitted 2014-02-19; First posted 2014-03-04 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Clinical Isolated Syndrome (CIS); Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- interferon beta-1a: 30 μg intramuscularly once a week using an injection device (Avonex Pen).
  Interventions: Device: interferon beta-1a

INTERVENTIONS:
Device: interferon beta-1a — Administered as specified in the treatment arm
  Other Names: BG9418; Avonex Pen; Avonex

SUMMARY:
To evaluate treatment tolerability, adherence and quality of life (QoL) over 1 year in MS (Multiple Sclerosis) participants who have been switched - due to persistent tolerability issues, particularly injection problems - from a subcutaneous injectable disease-modifying treatment (DMT) given several times a week (Rebif, Betaferon or Copaxone) to once weekly Avonex 30 μg given intra-muscularly. Avonex will be applied by the injection device Avonex Pen.

ELIGIBILITY:
Key Inclusion Criteria:

* Continuous treatment with Rebif, Betaferon or Copaxone over at least the past year.
* Injections site tolerability issues documented in medical records or by a nurse at inclusion.
* Clinically stable (free from relapses and 6-month confirmed disability progression for at least 6 months) while on therapy.
* Documented neurological history at least for the year prior to study entry.
* Qualification for Avonex® (Avonex Pen) according to the approved indication (Clinical Isolated Syndrome) or Relapsing Remitting Multiple Sclerosis (RRMS).
* Acceptance of magnetic resonance imaging.

Key Exclusion Criteria:

* Patients who have previously entered this study.
* Treatment with Avonex during the 12 months prior to the study.
* One or more relapses and/or 6-month confirmed disability progression during the 6 months prior to the study.
* Patient on Betaferon with Neutralizing Antibodies (NAbs) more than 400 TRU (tenfold reduction units) and patients on Rebif with NAbs with more than 100 TRU.
* Secondary progressive multiple sclerosis.
* Primary progressive multiple sclerosis.
* Pregnancy or breast feeding.
* History of severe depression or attempted suicide or current suicidal ideation.
* Medical or psychiatric conditions that compromise the ability to give informed consent, to comply with the protocol, or to complete the study.
* Uncontrolled seizure disorder.
* Myopathy or clinically significant liver disease.
* Inability, in the opinion of the principal investigator or staff, to comply with protocol requirements for the duration of the study.
* Known hypersensitivity to interferon-beta or other human proteins including albumin.
* A history of drug abuse in the 6 months prior to screening.
* Treatment with any of the following in the 30 days before day 1: systemic corticosteroids, ACTH, or other investigational drugs.
* Participation in any other study involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment by participating clinicians in Switzerland and Czech Republic.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to month 4 in injection site tolerability as measured on a composite visual analogue scale (VAS) score ranging from 0-100 | Up to 4 months

SECONDARY OUTCOMES:
Change from baseline to month 12 in injection site tolerability as measured on a composite VAS score | Up to 12 months
Change from baseline in the VAS score of systemic tolerability | Up to 12 months
The percentage of participants still on Avonex Pen | Up to 12 months
Quality of Life as assessed by the change in Short Form (SF) Health Survey, SF-36 scores | Up to 12 months
  The SF-36 is a short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
The percentage of missed injections | Up to 12 months
Change in Fatigue Scale for Motor and Cognitive functions (FSMC) score | Up to 12 months
  Fatigue is rated using the self-administered FSMC questionnaire that includes ten questions that relate to motor fatigue and ten to cognitive fatigue. Higher scores indicate higher fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- Czechia (6):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Teplice
- Switzerland (5):
  - Research Site, Biel/Bienne
  - Research Site, Langenthal
  - Research Site, Lugano
  - Research Site, Sion
  - Research Site, Wil